CLINICAL TRIAL: NCT05981183
Title: A Single Center Pilot Study on the Use of a Transcutaneous Auricular Vagus Nerve Stimulation Device in CKD Population
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation Device in CKD Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-00778
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention A (Experimental): Participants will receive 15 minutes of taVNS after an initial 15 minute rest-period and a 15 minute baseline measurement period. For participants assigned to Intervention A, the pulse width = 250 μs, and frequency = 50 Hz.
  Interventions: Device: Transcutaneous electrical nerve stimulation unit (TENS)
- Intervention B (Experimental): Participants will receive 15 minutes of taVNS after an initial 15 minute rest-period and a 15 minute baseline measurement period. For participants assigned to Intervention B, the pulse width = 300 μs, frequency = 25 Hz.
  Interventions: Device: Transcutaneous electrical nerve stimulation unit (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation unit (TENS) — The TENS unit will be applied to participants' right ear at the cymba conchae. The dose is dependent on which arm (Intervention A or Intervention B) the participant is assigned to. Participants will undergo 15 minutes of vagal nerve stimulation.
  Other Names: TENS Device 7000

SUMMARY:
The purpose of this pilot interventional study is to collect preliminary data on the application of a transcutaneous auricular vagal nerve stimulation (taVNS) device in patients with chronic kidney disease (CKD). This data will enhance understanding of the short-term safety, tolerability and effects of this novel therapeutic approach in the setting of CKD. The primary aims are to investigate the feasibility of the protocol and generate preliminary signals of efficacy and tolerability for two different doses of vagal nerve stimulation. The pilot estimates will be used to design a larger scale study that may lead to potentially targeted interventions to reduce cardiovascular (CV) mortality in the CKD population.

ELIGIBILITY:
Inclusion Criteria:

• Individual 18-80 years of age with CKD stage 3-5 (eGFR <60 mL/min/1.73m2) on most recent outpatient labs.

Exclusion Criteria:

* Pacemaker dependent
* Prisoners
* Pregnant women. A pregnancy test will be offered if a subject is concerned about being pregnant.
* Not capable of informed consent
* Know autonomic function disorder (e.g. Parkinson's disease with autonomic dysfunction)
* ICD or PPM precluding assessment of heart rate variability (e.g. chronic atrial fibrillation)
* Recent myocardial infarction (4 weeks or less)
* Maintenance dialysis
* Epilepsy
* Patients on labetalol (labetalol will interfere with catecholamine measurements)
* Patients with diabetes
* At least 50% of cohort must not be on beta blockers. This will help to distinguish the confounding effects of beta blockers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) at Baseline | Day 1 (15 minutes prior to administration of intervention)
  HRV is the variation in the time interval between heartbeats.
HRV at Post-Intervention | Day 1 (15 minutes Post-Intervention)
  HRV is the variation in the time interval between heartbeats.

SECONDARY OUTCOMES:
Percentage of Participants with at least a 20% change in HRV from baseline to post-intervention | Day 1 (Up to 15 Minutes Post-Intervention)
  The percentage of participants whose measured HRV changes by more than 20% from the baseline measurement to the post-intervention measurement.
Blood Pressure at Baseline | Day 1 (15 minutes prior to administration of intervention)
  Blood pressure measured continuously for 15 minutes prior to intervention.
Blood Pressure at Post-Intervention | Day 1 (15 minutes Post-Intervention)
  Blood pressure measured continuously for 15 minutes post-intervention.
Spontaneous Baroreceptor Sensitivity (BRS) at Baseline | Day 1 (15 minutes prior to administration of intervention)
  Spontaneous BRS is defined as the change in interbeat interval (IBI) in milliseconds per unit change in blood pressure.
Spontaneous BRS at Post-Intervention | Day 1 (15 minutes Post-Intervention)
  Spontaneous BRS is defined as the change in interbeat interval (IBI) in milliseconds per unit change in blood pressure.
Heart Rate at Baseline | Day 1 (15 minutes prior to administration of intervention)
Heart Rate at Post-Intervention | Day 1 (15 minutes Post-Intervention)

CONTACTS AND LOCATIONS:
Overall Officials: David Charytan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: David.Charytan@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to David.Charytan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.